CLINICAL TRIAL: NCT06292988
Title: Predective Factors for Tumor Aggressiveness in Medullary Thyroid Cancer
Brief Title: Predictive Factors for Medullary Thyroid Cancer Aggressiveness
Acronym: MYELO
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Associate Professor, Aristotle University Of Thessaloniki
Other Study IDs: MYELO
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-03

CONDITIONS: Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Total Thyroidectomy — Total thyroidectomy

SUMMARY:
This study is a retrospective study trying to find the predictive factors for medullary thyroid aggressiveness in terms of tumor metastasis and patients' survival.

DETAILED DESCRIPTION:
This study is a retrospective study trying to find the predictive factors for medullary thyroid aggressiveness in terms of tumor metastasis and patients' survival. The predictive factors included in this study are central and lateral compartment lymph node metastases as well as distant metastasis up to 1 year postoperatively, while biochemical predictors (meaning ratios such as lymphocyte to monocyte ratio etc and CEA and calcitonin drop levels) and histological predictors (such as nuclear atypia, amyloid, immunohistochemistry, desmoplasia) are included as secondary outcomes. In this study , patients >18 years old that underwent surgery for medullary thyroid cancer (total thyroidectomy, completion thyroidectomy) +/- central/lateral neck dissection) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent thyroidectomy for medullary thyroid cancer (total thyroidectomy, completion thyroidectomy) +/- central/lateral neck dissection

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years old who underwent surgery for medullary thyroid cancer are enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Central lymph node metastasis | Number of lymph node Metastasis found in preoperative imaging studies or up to 1 year postoperatively
  Central neck compartment lymph node metastasis
Lateral lymph node metastasis | Number of lymph node Metastasis found in preoperative imaging studies or up to 1 year postoperatively
  Lateral neck compartment lymph node metastasis
Distant metastasis | Number of distant Metastasis found in preoperative imaging studies or up to 1 year postoperatively
  Liver and lung metastasis

SECONDARY OUTCOMES:
Nuclear atypia as histological predictor of aggressiveness | The pathology report is held immediately after surgery
  nuclear atypia
Amyloid as histological predictor of aggressiveness | The pathology report is held immediately after surgery
  amyloid
Immunohistochemistry as histological predictor of aggressiveness | The pathology report is held immediately after surgery
  immunohistochemistry
Desmoplasia as histological predictor of aggressiveness | The pathology report is held immediately after surgery
  desmoplasia
CEA as Biochemical predictor of aggressiveness | pre and postoperative laboratory exams up to 1 year postoperatively
  Carcinoembryonic antigen (CEA) preoperatively and up to 1 year postoperatively
Calcitonin as Biochemical predictor of aggressiveness | pre and postoperative laboratory exams up to 1 year postoperatively
  calcitonin levels preoperatively and up to 1 year postoperatively
White blood cell as Biochemical predictor of aggressiveness | pre and postoperative laboratory exams up to 1 year postoperatively
  white blood cell count
Platelet count as Biochemical predictor of aggressiveness | pre and postoperative laboratory exams up to 1 year postoperatively
  platelet count
CEA drop as Biochemical cure marker | up to 1 year postoperatively
  CEA drop levels
Calcitonin drop as Biochemical cure marker | up to 1 year postoperatively
  calcitonin drop levels

CONTACTS AND LOCATIONS:
Overall Officials: Theodossis Papavramidis, Prof, Principal Investigator — 1st Propedeutic Department of Surgery, AHEPA University Hospital of Thessaloniki, Greece
Locations (46):
- Oregon Health & Science University, Oregon, Oregon City, Oregon, United States
- Department of Surgery, Saint John of God Hospital, Salzburg, Austria, Salzburg, Austria
- Saint Luc, University Clouvain, Belgium, Brussels, Belgium
- Head and Neck Surgery Department, Hospital Ana Nery, Santa Cruz do Sul, Brazil, Santa Cruz do Sul, Brazil
- University Clinic of Surgery, University Hospital "Lozenec", Sofia, Bulgaria
- Chinese University of Hong Kong, Hong Kong, China
- Head and Neck Department Oncologos del Occidente, Universidad de Caldas, Manizales, Colombia, Manizales, Colombia
- the University Hospital Center Sestre milosrdnice, Zagreb, Croatia, Department of Otorhinolaryngology and Head and Neck Surgery, Zagreb, Croatia
- France (2):
  - Head and Neck Surgery, Brest University Hospital, Brest, France, Brest
  - The University Hospital of Poitiers, France, Poitiers
- Greece (5):
  - Thyroid Surgery Clinic IKE, Athens, Greece, Athens
  - ENT Department University Hospital of Larissa, Larissa
  - Department of Surgery, General University Hospital of Patras, Pátrai
  - Aristotle University of Thessaloniki, Thessaloniki
  - Gennimatas General Hospital, Thessaloniki
- India (5):
  - Department of ENT-Head and Neck Surgery, All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar
  - KMCH and KMCH Comprehensive Cancer Center, Coimbatore
  - Department of Endocrine and Breast Surgery at Sanjay Gandhi Post Graduate Institute of Medical Sciences, Madurai
  - Department of Surgery, Maulana Azad Medical College & Lok Nayak Hospital, New Delhi
  - Endocrine and Metabolic Surgery, Bhargav Endocrine Hospital, Vijayawada, India, Vijayawada
- University of Sulaimani | UNIVSUL ,Department of Surgery, Kurdistan, Erbil, Iraq
- Italy (6):
  - ASL VCO - San Biagio Hospital - Domodossola (VB) - Italy, Domodossola
  - Dipartimento di Scienze Chirurgiche (DISC), University of Genoa, Italy, Genoa
  - Asst Santi Paolo e Carlo - Ospedale Polo Universitario San Paolo, Milan, Italy, Milan
  - UOC Chirurgia Endocrina e Metabolica, Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Department of Medical and Surgical Sciences, University of Trieste, Cattinara Teaching Hospital, Trieste, Italy, Trieste
  - Department of Surgery and Oncology, Endocrine Surgery Unit, Verona University Hospital, Verona
- Hashemite University of Zarqa, Zarqa, Jordan
- Hepatobiliairy and endocrine surgery, Ibn Sina Hospital, Medical School of Medecine Rabat, Mohamed Vth University of Rabat Morocco, Marrakesh, Morocco
- Division of General, Endocrine and Transplant Surgery, Medical University of Gdańsk, Gdansk, Poland
- Surgical Oncology Clinic, Institute for Oncology and Radiology of Serbia, Medical School, University of Belgrade, Belgrade, Serbia
- Slovakia (2):
  - Comenius University in Bratislava, Department of Paediatric Surgery, National Institute of Children's Diseases, Bratislava
  - Department of oncological surgery, St. Elisabeth cancer Institute, Bratislava
- Spain (4):
  - Hospital Clinic (Barcelona, Spain), Barcelona
  - Universitaria de Cordoba, Córdoba
  - Hospital Regional de Málaga, Málaga
  - Department of General and Digestive Surgery, Division of Endocrine Surgery, Complexo Hospitalario Universitario de Vigo, Vigo, Spain, Vigo
- Switzerland (2):
  - Bern University Hospital, Bern
  - Geneva University Hospital, Geneva
- Division of Endocrinology and Metabolism Department of Medicine Faculty of Medicine Ramathibodi Hospital Mahidol University Bangkok, Thailand, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Ankara University Faculty of Medicine, Department of Endocrine Surgery, Ankara
  - Acibadem MAA University, Istanbul
  - Cerrahpasa medical faculty endocrine surgery department, Istanbul
  - Department of Endocrin Pathology Unit, University of Health Sciences, Faculty of Medicine, Bakırköy Dr Sadi Konuk Training and Research Hospital, Istanbul, Turkey, Istanbul
- Endocrine surgeon-consultant, International medical center "CITIDOCTOR", Kyiv, Ukraine
- Department of Radiology, Thien Hanh Hospital, Buon Ma Thuot, Vietnam, Việt Trì, Vietnam

IPD SHARING:
Plan to Share IPD: No